CLINICAL TRIAL: NCT04875650
Title: Comparison of Physics Forceps and Conventional Forceps in Extraction of Mandibular Molars: A Double-Blinded Randomized Controlled Trial
Brief Title: Physics Forceps vs Conventional Forceps in Extraction of Mandibular Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melaka Manipal Medical College (Other)
Responsible Party: Principal Investigator, Auric Bhattacharya, Principal Investigator, Associate Professor, Melaka Manipal Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMMC/FOD/AR/B8/E C-2020 (01)
Record Dates: First submitted 2021-04-28; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Tooth Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physics Forceps (Experimental)
  Interventions: Procedure: Extraction of Mandibular Molar using Physics Forceps
- Conventional Forcep (Other)
  Interventions: Procedure: Extraction of Mandibular Molar using Conventional Forceps

INTERVENTIONS:
Procedure: Extraction of Mandibular Molar using Physics Forceps — Extraction of mandibular molars using physics forceps
  Arms: Physics Forceps
Procedure: Extraction of Mandibular Molar using Conventional Forceps — Extraction of mandibular molars using conventional forceps
  Arms: Conventional Forcep

SUMMARY:
Our study compared two different forceps for extraction of mandibular molars, the conventional extraction forceps and the Physics forceps. We assesed the relative pain score, patient satisfaction, success of extraction, incidence of alveolar plate fracture and soft tissue healing; post extraction. Our results found statistical significance in comparison of both forceps under relative pain score, patient satisfaction and soft tissue healing post extraction.

DETAILED DESCRIPTION:
Abstract

* INTRODUCTION/ BACKGROUND Tooth extractions are commonly done with conventional forceps. Recent advances like physics forceps help in atraumatic extractions by preserving the buccal plate, having less pain and better gingival healing. The buccal portion of the forceps is a plastic covered bumper which prevents reflection of buccal gingiva and buccal plate fracture. This is the first such comparison study to measure gingival healing in mandibular molar region with D2 bone quality.
* OBJECTIVE To compare the efficacy of Physics Forceps and Conventional Forceps in extraction of mandibular molars by randomly dividing the patients in two groups. The efficacy is determined by comparing the success of extraction, relative pain score, incidence of alveolar fracture, patient satisfaction and soft tissue healing on 3rd post-operative day.
* METHODOLOGY Patients who were indicated for extraction were included in the study. They were divided into two groups of 10 by double blinded randomization. Local Anesthesia was administered and the extraction was carried out using either Physics or Conventional forceps. Post extraction, the pain score was assessed using the VAS. Along with these, the gingival healing, success of extraction and alveolar plate fracture was assessed by the subject expert on the 3rd day post-operative day.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-55 years
* Mandibular molar teeth indicated for extractions with gingival index 1.

Exclusion Criteria:

* Patients with uncontrolled systemic diseases, that compromise dental extraction
* Mandibular 3rd Molars
* Grade 2 and 3 mobile teeth
* Grossly decayed mandibular molars

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Relative Pain Score | Day 1
  Use of a Visual Analogue Scale with 0 meaning no pain and 100 meaning severe pain
Soft Tissue Healing Post Extraction | Day 3
  Soft Tissue Healing Index by Landry et al.
Patient Satisfaction | Day 1
  4 point likert scale where 1 is very dissatisfied and 4 is very satisfied
Success of Extraction | Day 1
  1 is Failure, 2 is limited success with osteotomy, 3 is limited success with root fracture, 4 is limited success with apical fracture and 5 is complete success
Incidence of Alveolar Bone Fracture | Day 1
  Fracture 1 and No fracture 0

CONTACTS AND LOCATIONS:
Overall Officials: Auric Bhattacharya, BDS, MDS, FICOI, MFDS, RCPS, Principal Investigator — Melaka Manipal Medical College
Locations (1):
- Melaka Manipal Medical College, Malacca, Malaysia